CLINICAL TRIAL: NCT02273401
Title: A Randomised, Double-blind, Placebo-controlled (Within Dose Groups) Study to Assess Safety, Tolerability and Pharmacokinetics of Single Rising Inhaled Doses (0.5 μg to 70 μg Administered With the Respimat®) of BI 11054 CL in Healthy Male Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Single Rising Inhaled Doses of BI 11054 CL Administered With the Respimat® in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1250.1
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- BI 11054 CL (Experimental)
  Interventions: Drug: BI 11054 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 11054 CL
  Arms: BI 11054 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate safety, tolerability, and pharmacokinetics of BI 11054

ELIGIBILITY:
Inclusion Criteria:

* Healthy male based upon a complete medical history, including the physical examination, regarding vital signs (BP, PR), 12-lead ECG measurement, and clinical laboratory tests. There is no finding deviating from normal and of clinical relevance. There is no evidence of a clinically relevant concomitant disease.
* Age ≥21 and ≤50 years
* Body mass index (BMI) ≥18.5 and <30 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR, and ECG measurements) deviating from normal and of clinical relevance
* Evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to the drug or its excipients) as judged clinically relevant by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to randomisation
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to randomisation
* Participation in another trial with an investigational drug within 2 months prior to randomisation
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days as judged by the investigator
* Alcohol abuse (more than 40 g alcohol a day)
* Drug abuse
* Blood donation (more than 100 mL blood within 4 weeks prior to randomisation or during the trial)
* Excessive physical activities within 1 week prior to randomisation or during the trial
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of the study centre

The following exclusion criteria are specific for this study due to the known class side effect profile of ß2-mimetics:

* Asthma or history of pulmonary hyperreactivity
* Hyperthyrosis
* Allergic rhinitis in need of treatment
* Clinically relevant cardiac arrhythmia
* Paroxysmal tachycardia (>100 beats per minute)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with clinically significant findings in physical examination | up to 18 days after drug administration
Number of subjects with clinically significant findings in vital signs | up to 18 days after drug administration
  blood pressure (BP), pulse rate (PR), respiratory rate (RR)
Number of subjects with clinically significant findings in orthostasis tests | up to 24 hours after drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 18 days after drug administration
Number of subjects with clinically significant findings in additional safety laboratory tests | up to 24 hours after drug administration
  cyclic adenosine monophosphate (cAMP) and potassium
Number of subjects with clinically significant changes in body temperature | up to 24 hours after drug administration
Number of subjects with clinically significant findings in electrocardiogram (ECG) | up to 18 days after drug administration
Number of subjects with adverse events | up to 18 days after drug administration
Number of subjects with findings of oropharyngeal inspection | up to 24 hours after drug administration
Number of subjects with findings of pulmonary auscultation | up to 24 hours after drug administration
Airway resistance (Raw) | up to 24 hours after drug administration
  measured by body plethysmography
Global tolerability assessed by investigator on a 4-point scale | up to 18 days after drug administration

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 96 hours
tmax (time from dosing to maximum measured concentration) | up to 96 hours
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable analyte plasma concentration) | up to 96 hours
AUCt1-t2 (area under the concentration-time curve of the analyte in plasma over the time interval from time t1 to time t2) | up to 96 hours
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 96 hours
%AUCtz-∞ (percentage of the AUCtz-∞ that is obtained by extrapolation) | up to 96 hours
λz (terminal rate constant in plasma) | up to 96 hours
t1/2 (terminal half-life of the analyte in plasma) | up to 96 hours
MRTih (mean residence time of the analyte in the body after inhalation) | up to 96 hours
CL/F (apparent clearance of the analyte in plasma after extravascular administration) | up to 96 hours
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 96 hours
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | up to 96 hours
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 96 hours
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 96 hours